CLINICAL TRIAL: NCT01032915
Title: A 24 Week Multi-center, Randomized, Double-masked, Placebo Controlled, Dose-ranging Phase III Study of AIN457 Versus Placebo for Maintaining Uveitis Suppression When Reducing Systemic Immunosuppression in Patients With Quiescent, Non-infectious Intermediate, Posterior or Panuveitis.
Brief Title: Safety and Efficacy of AIN457 in Patients With Quiescent Non-infectious Uveitis
Acronym: ENDURE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Results of a planned interim analysis did not show significant effects for any of the 3 AIN dose regimens versus placebo on any primary or secondary endpoint
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457C2301; 2009-014835-19 (EudraCT Number)
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Results first posted 2015-11-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-10

CONDITIONS: Non-infectious Uveitis
Keywords: Quiescent uveitis; intermediate uveitis; panuveitis; posterior uveitis; uveitis
MeSH Terms: conditions — Uveitis, Intermediate; Panuveitis; Uveitis, Posterior; Uveitis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AIN457 300mg s.c weekly for 3 weeks (Experimental): AIN457 300mg s.c weekly for 3 weeks then every 2 weeks
  Interventions: Biological: AIN457
- AIN457 300mg s.c at baseline and Week 2 (Experimental): AIN457 300mg s.c at baseline and Week 2 then every 4 weeks
  Interventions: Biological: AIN457
- AIN457 150mg s.c at baseline and Week 2 (Experimental): AIN457 150mg s.c at baseline and Week 2 then every 4 weeks
  Interventions: Biological: AIN457
- Placebo s.c weekly for 3 weeks (Placebo Comparator): Placebo s.c weekly for 3 weeks then every 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: AIN457 — AIN457 300mg s.c weekly for 3 weeks then every 2 weeks
  Arms: AIN457 300mg s.c weekly for 3 weeks
Biological: AIN457 — AIN457 300mg s.c at baseline and Week 2 then every 4 weeks
  Arms: AIN457 300mg s.c at baseline and Week 2
Biological: AIN457 — AIN457 150mg s.c at baseline and Week 2 then every 4 weeks
  Arms: AIN457 150mg s.c at baseline and Week 2
Drug: Placebo — Placebo s.c weekly for 3 weeks then every 2 weeks
  Arms: Placebo s.c weekly for 3 weeks

SUMMARY:
This study will assess the safety and efficacy of AIN457 as adjunctive therapy for the treatment of intermediate uveitis, posterior uveitis, or panuveitis requiring systemic immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with quiescent chronic, non-infectious intermediate uveitis, posterior uveitis or panuveitis as evidenced by <1+ anterior chamber cell grade and <1+ vitreous haze in both eyes for at least 6 weeks prior to screening.
* Requirement for either of the following immunosuppressive therapies at any time within the past 3 months for the treatment or prevention of uveitis which must not have been increased within the 6 weeks prior to screening:

Prednisone or equivalent ≥10 mg daily.

≥1 periocular injection or ≥1 intravitreal corticosteroid injection (i.e. triamcinolone) in the study eye within the past 6 months (the last injection must not have been given 6 weeks prior to screening.)

Treatment with either cyclosporine, tacrolimus, azathioprine, mycophenolate mofetil, mycophenolic acid, methotrexate as monotherapy or in combination with or without steroids. (Patients treated with chlorambucil or cyclophosphamide within the past 5 years are ineligible for the study.)

Patients not meeting the above specified criteria for immunosuppressive therapies are eligible for enrollment if they are intolerant to systemic immunosuppressive therapy as determined by the study investigator.

Exclusion Criteria:

Ocular concomitant conditions/disease

* Patients with a primary diagnosis of Behcet's disease, anterior uveitis or any intermediate uveitis, posterior uveitis or panuveitis in which the manifestation(s) of the active intraocular inflammatory disease may spontaneously resolve or that are not characterized by the presence of either anterior chamber cells or vitritis (vitreous cell and haze) such as the white dot retino-choroidopathies (i.e. Punctate inner choroidopathy (PIC), acute zonal occult outer retinopathy (AZOOR.)
* Patients with active, non-infectious intermediate, posterior or panuveitis in one or both eyes (≥1+ anterior chamber cells and /or ≥1+ vitreous haze.)
* Patients receiving or that may require corticosteroids (prednisone or equivalent) ≥1 mg/kg/day to maintain quiescence of their intraocular inflammation.

Ocular treatments

* Treatment with intravitreal anti-VEGF agents administered to the study eye within 3 months prior to screening.
* Treatment with fluocinolone acetonide implant (Retisert®) in the study eye within the last 3 years, or dexamethasone intravitreal implant and any other investigational corticosteroid implants in the study eye within the last 6 months.
* Intraocular surgery or laser photocoagulation in the study eye within the last 6 weeks prior to screening except for a diagnostic vitreous or aqueous tap with a small-gauge needle.

Systemic conditions or treatments

* Any systemic biologic therapy (e.g. interferon, infliximab, daclizumab, etanercept, or adalimumab) given intravenously or subcutaneously within 3 months prior to screening. No biologic therapy other than the investigational study treatment will be allowed during the course of the clinical trial.
* Any prior treatment with systemic alkylating agents (cyclophosphamide, chlorambucil) within the past 5 years prior to screening.
* Treatment with any live or live-attenuated vaccine (including vaccine for varicella-zoster or measles) within 2 months prior to screening. No treatment with live or live-attenuated vaccines will be allowed during the course of the clinical trial.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (82):
- United States (24):
  - Sall Research Medical Center, Artesia, California
  - Novartis Investigative Site, Artesia, California
  - Novartis Investigative Site, Beverly Hills, California
  - Retina-Vitreous Assoc. Medical Group, Beverly Hills, California
  - Emory University, Atlanta, Georgia
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Louisville, Kentucky
  - University of Louisville Opthamology, Louisville, Kentucky
  - Novartis Investigative Site, Baltimore, Maryland
  - The Wilmer Eye Institute, Baltimore, Maryland
  - Massachusets Eye Research and Surgery Institution (MERSI), Cambridge, Massachusetts
  - Novartis Investigative Site, Cambridge, Massachusetts
  - Novartis Investigative Site, Teaneck, New Jersey
  - The Cornea and Laser Institute and UMDNJ, Teaneck, New Jersey
  - Charlotte Eye, Ear, Nose, and Throat Associates, Belmont, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Portland, Oregon
  - OHSU, Casey Eye Institute, Portland, Oregon
  - Novartis Investigative Site, Arlington, Texas
  - Texas Retina Associates, Arlington, Texas
  - Houston Eye Associates, Houston, Texas
  - Novartis Investigative Site, Houston, Texas
  - University of Washington, Seattle, Washington
  - Novartis Investigative Site, Seattle, Washington
- Brazil (3):
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, São Paulo
- Germany (8):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Tübingen
- India (10):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Chandigarh
  - Novartis Investigative Site, Chennai
  - Novartis Investigative SIte, Coimbatore
  - Novartis Investigative Site, Kolkata
  - Novartis Investigative Site, Madurai
  - Novartis Investigative Site, New Delhi
- Israel (4):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (7):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Ancona
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Parma
  - Novartis Investigative Site, Roma
- Spain (10):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Barakaldo
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Santiago de Compostela
  - Novartis Investigative Site, Valencia
- Switzerland (8):
  - Novartis Investigative Site, Lausanne, CHE
  - Novartis Investigative Site, Lausanne, Switzerland
  - Novartis Investigative Site, Zurich, Switzerland
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Lucerne
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Zurich
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Fatih / Istanbul
  - Novartis Investigative Site, Istanbul
- United Kingdom (5):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, York

REFERENCES:
- [Derived] Dick AD, Tugal-Tutkun I, Foster S, Zierhut M, Melissa Liew SH, Bezlyak V, Androudi S. Secukinumab in the treatment of noninfectious uveitis: results of three randomized, controlled clinical trials. Ophthalmology. 2013 Apr;120(4):777-87. doi: 10.1016/j.ophtha.2012.09.040. Epub 2013 Jan 3. PMID 23290985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2010 and March 2011, 125 patients were randomized from 51 centers in 9 countries (United States, Germany, Switzerland, India, Spain, United Kingdom, Israel, Brazil and Italy). Recruitment did not reach the target of 340 patients due to early termination of the study.
Groups:
- AIN457 300mg s.c Every 2 Weeks: AIN457 300mg s.c weekly for 3 weeks, then every 2 weeks
- AIN457 300mg s.c Every 4 Weeks: AIN457 300mg s.c at baseline and Week 2, then every 4 weeks
- AIN457 150mg s.c Every 4 Weeks: AIN457 150mg s.c at baseline and Week 2, then every 4 weeks
- Placebo s.c Every 2 Weeks: Placebo s.c weekly for 3 weeks, then every 2 weeks
Period: Overall Study
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks
Started | 29 | 31 | 31 | 34
Completed | 21 | 20 | 24 | 27
Not Completed | 8 | 11 | 7 | 7
Not completed — Adverse Event | 2 | 2 | 1 | 1
Not completed — Abnormal test procedure result | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1 | 1
Not completed — Administrative reasons | 5 | 6 | 4 | 4
Not completed — Protocol Violation | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Set: This set included all randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks | Total
Number analyzed (Participants) | 29 | 31 | 31 | 34 | 125
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.2 (14.29) | 49.2 (11.14) | 47.7 (13.5) | 47.3 (15.46) | 47.6 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 20 | 18 | 71
  Male | 12 | 15 | 11 | 16 | 54

OUTCOME MEASURES:

1. Primary Outcome: Time to First Recurrence in Any Eye of Active Intermediate, Posterior, or Panuveitis From Baseline
Description: Kaplan-Meier estimates for the time to the first recurrence in any eye of active intermediate, posterior, or panuveitis from baselineRecurrence of active intermediate, posterior, or panuveitis defined by either: ≥ 2 step increase in vitreous haze with or without an increase in anterior chamber cell grade or decrease in best corrected visual acuity of ≥ 10 ETDRS letters
Time Frame: Baseline to 24 weeks
Population: Full Analysis Set (FAS): all randomized patients who received at least one dose of study drug and have at least one post-baseline assessment for the primary efficacy parameter or any of its components. Following the intent-to-treat principle, patients were analyzed according to the treatment they are assigned to at randomization.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks
Number analyzed (Participants) | 29 | 31 | 31 | 33
Days | NA [NA to NA] — Not estimable due to low number of events | NA [87 to NA] — Not estimable due to low number of events | 178 [178 to NA] — Not estimable due to low number of events | NA [170 to NA] — Not estimable due to low number of events

2. Secondary Outcome: Change (Reduction) From Baseline in Composite Immunosuppressive Medication Score (IMS) From Baseline to 24 Weeks
Description: Participants could have received up to 5 immunosuppresive agents (prednisone, cyclosporine, azathioprine, methotrexate, mycophenolate). Immunosuppressive Medication Score (IMS) is a combined, single numeric score derived on basis of total daily dose of specific immunosuppressive agents / unit body weight, ranged on a scale from 0-9 for the total daily dose in mg per kg. Patients receiving multiple medications, the sum of the grading scores for each drug was used to calculate a total immunosuppression score at each visit. The total IMS is the sum of scores derived from the agents included into the score, and ranged from 0 to 55. Treatment groups compared using analysis of covariance with treatment & baseline IMS as covariate, where the lower IMS (or its reduction from baseline) showed better clinical outcome
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks
Number analyzed (Participants) | 29 | 31 | 31 | 33
Score | -2.55 (3.22) | -2.81 (2.847) | -2.92 (2.874) | -2.13 (3.049)

3. Secondary Outcome: Mean Change in Best Corrected Visual Acuity From Baseline
Description: The Best Corrected Visual Acuity (BCVA) is tested using the Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity (VA) testing protocol. VA measurements are taken in a sitting position at an initial test distance of 4 meters using ETDRS charts. The overall BCVA score is calculated using the BCVA worksheet 0-100 letter score.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks
Number analyzed (Participants) | 29 | 31 | 31 | 33
Letters | 2.9 (4.86) | 1.8 (6.12) | 1.9 (4.46) | 1.4 (9.42)

4. Secondary Outcome: Mean Change in Vitreous Haze Grade From Baseline to 24 Weeks
Description: The changes in steps (0, 1, or >= 2) from previous visit for vitreous haze, where the score is evaluated based on NEI Vitreous Haze Grading Scale (0 -4). Vitreous haze was recorded as 0-clear; to 4+ as dense opacity obscuring the optic nerve head. A 1 step increase is defined as any of the following changes: 0-1, 0.5-1, 1-2, 2-3, 3-4. A 2 step increase is defined as any of the following changes: 0-2, 0.5-2, 1-3, 2-4. A recurrent episode of active intermediate, posterior or panuveitis was considered to be resolved, if the eye returns and maintains in a quiescent state (<1+ anterior chamber cell grade and <1+ vitreous haze) for at least 2 weeks
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks
Number analyzed (Participants) | 29 | 31 | 31 | 33
Score | 0.02 (0.295) | 0.03 (0.197) | 0.02 (0.232) | 0.2 (0.465)

ADVERSE EVENTS:
Description: Safety Analysis Set: The safety set consists of all patients who received at least one dose of study drug and have at least one post-baseline safety assessment. Patients were analyzed according to the treatment they actually received, regardless of study drug relationship, by system preferred term
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks
Serious Adverse Events (participants affected / at risk) | 2/29 | 1/31 | 0/31 | 1/33
Other Adverse Events (participants affected / at risk) | 14/29 | 17/31 | 19/31 | 14/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300mg s.c Every 2 Weeks (N=29) | AIN457 300mg s.c Every 4 Weeks (N=31) | AIN457 150mg s.c Every 4 Weeks (N=31) | Placebo s.c Every 2 Weeks (N=33)
Uveitis (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Mononeuropathy multiplex (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300mg s.c Every 2 Weeks (N=29) | AIN457 300mg s.c Every 4 Weeks (N=31) | AIN457 150mg s.c Every 4 Weeks (N=31) | Placebo s.c Every 2 Weeks (N=33)
Cataract subcapsular (Study eye) (Eye disorders) | 1 | 0 | 2 | 1
Conjunctivitis (Fellow eye) (Eye disorders) | 0 | 1 | 2 | 0
Dry eye (Fellow eye) (Eye disorders) | 0 | 2 | 1 | 0
Dry eye (Study eye) (Eye disorders) | 0 | 2 | 1 | 0
Macular oedema (Fellow eye) (Eye disorders) | 1 | 0 | 1 | 2
Vision blurred (Fellow eye) (Eye disorders) | 2 | 1 | 0 | 1
Vision blurred (Study eye) (Eye disorders) | 2 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 2
Asthenia (General disorders) | 0 | 0 | 2 | 1
Ear infection (Infections and infestations) | 1 | 2 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 2 | 0
Influenza (Infections and infestations) | 2 | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 2 | 4 | 3
Oral herpes (Infections and infestations) | 0 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 4
Headache (Nervous system disorders) | 5 | 4 | 2 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety